CLINICAL TRIAL: NCT02673242
Title: Inspiratory Muscle Training for Patients With Chronic Obstructive Pulmonary Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Bergen University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E16260
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Control (No Intervention): No treatment other than medical
- Intervention (Experimental): Inspiratory muscle training
  Interventions: Device: Threshold IMT Philips Respironics

INTERVENTIONS:
Device: Threshold IMT Philips Respironics — Inspiratory muscle training
  Arms: Intervention

SUMMARY:
This study is a randomized controlled trial with the aim of evaluating the effect of homebased inspiratory muscle training (IMT) for patients with COPD in Norway. The intervention group will train with threshold IMT for 6 weeks. The control group will not participate in any other training method or sham. Evaluation parameters are maximal inspiratory pressure, six minute walk test, COPD assessment test, modified Medical research council dyspnea scale and spirometry.

ELIGIBILITY:
Inclusion Criteria:

* COPD grade III-IV,
* Inhabitant of Hedmark (Løten, Våler, Åsnes, Hamar, Elverum)

Exclusion Criteria:

* Undergoing exercise based physical therapy treatment,
* not able to do IMT physically or mentally

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory pressure | 6 weeks

SECONDARY OUTCOMES:
Six minute walk test | 6 weeks
Modified Medical Research Council Dyspnea Scale | 6 weeks
COPD Assessment Test | 6 weeks
Spirometry | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sykehuset Innlandet Hospital Trust, Elverum, Norway

IPD SHARING:
Plan to Share IPD: No